CLINICAL TRIAL: NCT00915707
Title: Pathways Linking Reduced Sleep Duration and Quality to Obesity Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 14916B
Record Dates: First submitted 2009-06-03; First posted 2009-06-08 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Diabetes
Keywords: obesity; diabetes, risk; obesity, diabetes risk related to sleep
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — BaseLine dental cement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline (Experimental): Subjects are tested under normal sleep conditions for carbohydrate metabolism and appetite regulation.
  Interventions: Other: Baseline
- Sleep restriction (Experimental): Subjects are tested under sleep restriction for carbohydrate metabolism and appetite regulation.
  Interventions: Other: Sleep restriction
- Reduced sleep quality (Experimental): Subjects are tested under a poor sleep quality condition for carbohydrate metabolism and appetite regulation.
  Interventions: Other: Reduced Sleep Quality

INTERVENTIONS:
Other: Baseline — Subjects are allowed time in bed for sleep as their usual time at home.
  Arms: Baseline
Other: Sleep restriction — Subjects sleep is reduced to 4.5 hours in bed for 4 nights.
  Arms: Sleep restriction
Other: Reduced Sleep Quality — Subjects sleep quality is reduced for 4 nights.
  Arms: Reduced sleep quality

SUMMARY:
This study is designed to study the pathways through which short sleep duration or poor sleep quality can lead to an increased risk of developing diabetes and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight
* Healthy
* Normal sleep times

Exclusion Criteria:

* Sleep disorders
* Overweight
* Diabetes
* Other health conditions
* Excessive caffeine and alcohol intake
* Smoking

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Disposition Index reflecting Diabetes Risk as a result of decreased sleep duration and/or quality. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States